CLINICAL TRIAL: NCT03477578
Title: Freezing of Gait and Cognition: What Can we Learn From Cognition?
Brief Title: Freezing of Gait and Cognition
Acronym: FOG-As-PD
Status: Completed | Type: Observational
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Other Study IDs: FOG-As-PD
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Gait Disorder, Sensorimotor; Cognition Disorders; Parkinson Disease
MeSH Terms: conditions — Gait Disorders, Neurologic; Cognition Disorders; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FoG+: Parkinsonian patients with Freezing of Gait
  Interventions: Other: freezers; Other: non freezers
- FoG-: Parkinsonian patients withou Freezing of Gait
  Interventions: Other: freezers; Other: non freezers

INTERVENTIONS:
Other: freezers — neuropsychological evaluation
Other: non freezers — neuropsychological evaluation

SUMMARY:
The study was aimed to investigate the role of cognition n in FoG.

DETAILED DESCRIPTION:
Alteration of cortical circuits in PD leads to cognitive dysfunctions associated with the development of FoG.

The study was aimed to investigate the role of cognition in FoG.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease according to Gelb et al.

Exclusion Criteria:

* Any other neurological conditions other than PD

Age Groups: Child, Adult, Older Adult
Study Population: Parkinsonian patients with and without freezing of gait hospitalized at the Department of Parkinson's disease, Movement Disorders and Brain Injury Rehabilitation, "Moriggia-Pelascini" Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
UPDRS | 5 years
  Unified Parkinson's DIsease Rating Scale
MMSE | 5 years
  Mini-Mental State Examination
FAB | 5 years
  Frontal Behavioural Assessment
WCST | 5 years
  Wisconsin Card Sorting Test
TMT A-B | 5 years
  Trial Making Test A and B
Rey Auditory-Verbal Learning Test | 5 years
  RAVLT

SECONDARY OUTCOMES:
6MWT | 5 years
  Six-Minute Walk Test
TUG | 5 years
  Timed Up and Go Test

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — Department of Parkinson's disease, Movement Disorders and Brain Injury Rehabilitation, "Moriggia-Pelascini" Hospital - Via Pelascini, 3, 22015, Gravedona ed Uniti, Como, Italy
Locations (1):
- "Moriggia-Pelascini" Hospital, Gravedona Ed Uniti, CO, Italy

IPD SHARING:
Plan to Share IPD: No